CLINICAL TRIAL: NCT00031213
Title: Heavy Metals, Obesity and Cardiovascular Risk - Ancillary to Look AHEAD
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 992; R01HL070299 (NIH)
Record Dates: First submitted 2002-02-27; First posted 2002-02-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Diabetes Mellitus, Non-insulin Dependent; Cardiovascular Diseases; Obesity; Myocardial Infarction; Heart Diseases; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity; Myocardial Infarction; Heart Diseases; Diabetes Mellitus

SUMMARY:
To evaluate the relationship of baseline toenail chromium concentrations to weight loss, as well as the interaction between heavy metals and the beneficial effects of weight loss.

DETAILED DESCRIPTION:
BACKGROUND:

Heavy metals are a heterogeneous group of highly reactive substances, which may act as essential cofactors for physiologic processes and/or as toxic elements. Chromium, in particular, has been associated with obesity, diabetes, and weight loss. Other heavy metals have been associated with some of the consequences of obesity, including hypertension, hyperlipidemia, and cardiovascular disease. The Look AHEAD Study, a large randomized controlled trial of intensive lifestyle intervention for weight loss in obese patients with Type 2 diabetes mellitus, provides an excellent opportunity to address the impact of chromium on weight loss and diabetes control, as well as to assess the impact of other heavy metals on the physiologic consequences of weight loss.

The study is ancillary to the Look AHEAD clinical trial which is sponsored primarily by the National Institute of Diabetes and Digestive and Kidney Diseases and secondarily by the National Heart, Lung, and Blood Institute, the National Institute of Nursing Research, the Office of Research on Women's Health, the National Center on Minority Health and Health Disparities, and the Centers for Disease Control and Prevention. The Look AHEAD study is a multicenter, randomized clinical trial to examine the long-term effects of a lifestyle intervention designed to achieve and maintain weight loss in overweight diabetics.

DESIGN NARRATIVE:

This is an ancillary prospective observational study within the Look AHEAD trial. The ancillary study will collect toenail clippings from all participants (n = 5,000) at baseline and at the 1-year visit, and analyze a random subset of the toenails for their heavy metal content using instrumental neutron activation analysis. Toenails provide a time-integrated measure of heavy metal exposure, while instrumental neutron activation analysis provides the concentrations of about 50 heavy metals in the toenail samples, including chromium. This information will allow an evaluation of the relationship of baseline toenail chromium concentrations to weight loss, as well as the interaction between heavy metals and the beneficial effects of weight loss. The proposed study may provide, valuable insight into the determinants of the efficacy of weight loss interventions. In fact, the Look AHEAD trial, because of its size, may be one of the few studies in which these relationships can be measured reliably. In addition, the ancillary study will permit the setup of a specimen bank of toenails to be used in future case-cohort or nested case-control studies of the association of heavy metals with Look AHEAD endpoints, especially myocardial infarction and cardiovascular death.

ELIGIBILITY:
An estimated 5,000 obese diabetic subjects from the Look AHEAD clinical trial. There will be 2,500 women (50%) and 30% minorities.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliseo Guallar — Johns Hopkins University